CLINICAL TRIAL: NCT04988685
Title: SIROOP Registry - a Prospective Registry Study to Evaluate the Outcomes of Coronary Artery Disease Patients Treated with SIROlimus or Paclitaxel Eluting Balloon Catheters
Acronym: SIROOP
Status: Recruiting | Type: Observational
Sponsor: Luzerner Kantonsspital (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Matthias Bossard, Principal Co-Investigator, Luzerner Kantonsspital
Other Study IDs: 2021-00615
Record Dates: First submitted 2021-07-25; First posted 2021-08-03 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Coronary Arteriosclerosis; Coronary Artery Calcification; Stable Chronic Angina; Angina Pectoris; Angina, Stable; Angina, Unstable; Stent Thrombosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease; Coronary Restenosis; Angina, Stable; Angina Pectoris; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment: The project ́s main goal is to collect baseline, clinical and procedural data as well as to assess angiographic and clinical outcomes of CAD patients treated with contemporary DCBs.
  Interventions: Device: Sirolimus Eluting Balloon

INTERVENTIONS:
Device: Sirolimus Eluting Balloon — PTCA with either a Sirolimus eluting balloon or Paclitaxel eluting balloon
  Other Names: Paclitaxel Eluting Balloon

SUMMARY:
The purpose of the SIROOP Registry is to retrospectively and prospectively collect baseline, clinical and procedural characteristics of patients who have undergone PCI and are treated with either currently available sirolimus or paclitaxel coated DCBs (see Table 1), irrespective of clinical presentation as well as to prospectively collect data about their clinical outcomes. Outcomes will be compared in different clinical subgroups. The impact of current DCBs in different clinical settings and coronary artery lesions on cardiovascular outcomes will be assessed.

DETAILED DESCRIPTION:
Objectives in detail:

* To evaluate procedural success, efficacy, performance and clinical outcomes among various patient cohorts, who undergo PCI using currently available DCBs:

  1. Periprocedural outcomes/complications, which will be analyzed, include: final result (e.g. residual stenosis, TIMI flow), dissections, perforations, prevalence of thrombus (assessed by angiography and intravascular imaging)
  2. Short and long-term clinical outcomes of interest comprise among others: new MI, unstable angina (UA), target lesion failure, target vessel revascularization, target lesion failure/ revascularization, repeat hospitalization, new/worsening heart failure, cardiogenic shock, stroke, bleedings, cardiovascular death and all-cause death.
* To describe procedural and clinical performance of various DCB, either alone or in combination with other stent and coronary scaffold devices
* To identify optimal strategies for lesion preparation in cases treated with DCB
* To identify possible predictors for TLR after treatment with DCB
* To describe early and late angiographic and OCT-findings among coronary artery disease (CAD) patients treated with DCB and/or various metallic stent and scaffold devices
* To evaluate the impact of different antithrombotic regimens on patient's clinical outcomes
* To study procedural and clinical outcomes among CAD patients requiring hemodynamic support using mechanical devices.
* To describe economic implications (cost-effectiveness) of various interventional treatments for CAD.

ELIGIBILITY:
Inclusion Criteria:

* Subject >18 years of age
* Patients with significant acute or chronic coronary de-novo lesions or ISR lesions requiring treatment using PCI
* Treatment with at least one DCB (device choice at the operator's discretion) In case of a patient with lesions treated at different procedural time, lesions will be separately collected and documented
* Subjects must be willing to sign a patient informed consent (PIC) or must have signed the General Consent (GK).

Exclusion Criteria:

* Patient is <18 years of age
* Patient unwilling or unable to provide informed consent
* pregnancy and lactation
* Indication for surgical revascularization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This registry will recruit consecutive patients treated with either DCB alone or a hybrid strategy (metallic stent plus DCB). Ideally any patient treated with a DCB will be included in the present registry, either presenting with a de-novo coronary lesion (either elective or urgent procedure), with a ST or ISR.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of target lesion failure (TLF) and target lesion revascularization (TLR) | at 1 year

SECONDARY OUTCOMES:
Rate of combination of major adverse cardiac and cerebrovascular events (MACCE) (including new MI, TLR or cardiovascular death) | at 180 days, 1, 2 and 5 years
Rate of MACE | at 180 days, 1, 2 and 5 years
Rate of new MI (NSTEMI / STEMI) | at 180 days, 1, 2 and 5 years
Rate of TIA or stroke | at 180 days, 1, 2 and 5 years
Rate of acute vessel closure | at 180 days, 1, 2 and 5 years
Rate of stent thrombosis or ISR | at 180 days, 1, 2 and 5 years
Rate of target vessel revascularization (TVR) | at 180 days, 1, 2 and 5 years
Rate of target lesion revascularization (TLR) | at 180 days, 1, 2 and 5 years
Rate of target lesion failure (TLF) | at 180 days, 1, 2 and 5 years
Rate of ischemia driven TLR | at 180 days, 1, 2 and 5 years
Rate of all-cause death | at 180 days, 1, 2 and 5 years
Rate of cardiac death | at 180 days, 1, 2 and 5 years
Rate of all myocardial infarction and TV-MI | at 180 days, 1, 2 and 5 years
Rate of rehospitalization for recurrent angina | at 180 days, 1, 2 and 5 years
Rate of hospitalization for HF | at 180 days, 1, 2 and 5 years
Rate of rehospitalization for HF, resuscitated cardiac arrest or implantable cardioverter- defibrillator (ICD) implantation | at 180 days, 1, 2 and 5 years
Rate of bleeding events (access site or non-access site related) according to the BARC classification | at 180 days, 1, 2 and 5 years
Rate of vascular complications (according to VARC criteria) | at 180 days, 1, 2 and 5 years
Rate of cardiogenic shock | at 180 days, 1, 2 and 5 years
Rate of acute renal failure/ contrast-induced nephropathy (CIN) | at 180 days, 1, 2 and 5 years
Rate of new ventricular arrhythmias | at 180 days, 1, 2 and 5 years
Rate of major adverse limb events (MALE) | at 180 days, 1, 2 and 5 years
Rate of new York Heart Association (NYHA) class | at 180 days, 1, 2 and 5 years
Rate of angina according to Canadian Cardiovascular Society (CCS) Score | at 180 days, 1, 2 and 5 years
Rate of procedural success (final diameter stenosis < 30% without flow-limiting dissections) | at 180 days, 1, 2 and 5 years
Rate of periprocedural complications (e.g. coronary perforations, no-reflow) | at 180 days, 1, 2 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Florim Cuculi, MD, Principal Investigator — Luzerner Kantonsspital
Locations (1):
- Luzerner Heart Centre, Lucerne, Canton of Lucerne, Switzerland

REFERENCES:
- [Background] Cioffi GM, Madanchi M, Attinger-Toller A, Bossard M, Cuculi F. Pushing the Boundaries: Drug-Coated Balloons to Treat a Calcified and Thrombotic Lesion in Acute Coronary Syndrome. Am J Case Rep. 2022 Oct 5;23:e936950. doi: 10.12659/AJCR.936950. PMID 36196027
- [Background] Madanchi M, Cioffi GM, Attinger-Toller A, Seiler T, Somm S, Koch T, Tersalvi G, Wolfrum M, Moccetti F, Toggweiler S, Kobza R, Levine MB, Garcia-Garcia HM, Bossard M, Cuculi F. Metal free percutaneous coronary interventions in all-comers: First experience with a novel sirolimus-coated balloon. Cardiol J. 2022;29(6):906-916. doi: 10.5603/CJ.a2022.0106. Epub 2022 Nov 17. PMID 36385601
- [Background] Madanchi M, Attinger-Toller A, Gjergjizi V, Majcen I, Cioffi GM, Epper A, Gnan E, Koch T, Zhi Y, Cuculi F, Bossard M. Treatment of coronary lesions with a novel crystalline sirolimus-coated balloon. Front Cardiovasc Med. 2024 Feb 13;11:1316580. doi: 10.3389/fcvm.2024.1316580. eCollection 2024. PMID 38414923
- [Background] Madanchi M, Bossard M, Majcen I, Cioffi GM, Ferraro F, Gnan E, Gjergjizi V, Zhi Y, Bade V, Wolfrum M, Moccetti F, Toggweiler S, Attinger-Toller A, Cuculi F. Outcomes following coronary chronic total occlusion revascularization with drug-coated balloons. J Invasive Cardiol. 2024 Mar;36(3). doi: 10.25270/jic/23.00260. PMID 38441987